CLINICAL TRIAL: NCT00000349
Title: Infusion Laboratory: Protocol 5 (Flupenthixol)
Brief Title: Infusion Laboratory: Protocol 5 (Flupenthixol) - 14
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: NIDA-3-0010-14; Y01-3-0010-14
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2002-12

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Flupenthixol

INTERVENTIONS:
Drug: Flupenthixol

SUMMARY:
The purpose of this study is to evaluate clinical safety issues pertaining to flupenthixol, to cocaine, and to their interaction, and to determine how pretreatment with flupenthixol modifies the subjective as well as physiological effects of cocaine. Taken together, these relatively D-1 selective agents can help determine the extent to which DA-1 binding affects the reinforcing effects of stimulants.

ELIGIBILITY:
Inclusion Criteria:

M/F, ages 21-50. Meet DSM-IV criteria for cocaine dependence. Agree to conditions of the study and sign informed consent.

Exclusion Criteria:

Psychiatric disorder that requires medication therapy. History of seizures. Pregnant and/or nuring women. Dependence on ETOH or benzodiazepines or other sedative/hypnotics. Acute hepatitis. Other medical condtions that deem participation to be unsafe.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0

PRIMARY OUTCOMES:
Degree of drug craving
History, incidence and amount of drug use
Type and severity of stimulant withdrawal symptoms
Characterization of study population
Population incidence of symptoms of depression, po
Frequency and intensity of drug use and sexual beh
Evidence of change in neurophysiology and brain ac
Evidence of change in subjective responses to coca
Clinical physiological response to cocaine challen
Degree to which study medication influences change

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States